CLINICAL TRIAL: NCT05210972
Title: Severity of Newly Diagnosed Coronary Artery Disease in Patients With Newly Diagnosed Diabetes and Pre-diabetes: A Cohort Study in a Cardiac Center in Saudi Arabia
Brief Title: Coronary Artery Disease Severity in Newly Diagnosed Dysglycemia
Status: Completed | Type: Observational
Sponsor: Saud Al Babtain Cardiac Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SBCC-IRB-2021-06
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Dysglycemia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes: Patients with level of HbA1c ≥ 6.5%, or Fasting blood glucose (FBG) ≥126 mg/dL, or a random plasma glucose (RBG) ≥ 200 mg/dL in a patient with classic symptoms of hyperglycemia.
  In the absence of unequivocal hyperglycemia, diagnosis will be based on two abnormal test results, for FBG or RBG and HbA1c, from the same sample or in two separate test samples.
  Interventions: Radiation: Cardiac catheterization
- Prediabetes: HbA1c 5.7-6.4% or FBG 110 mg/dL to 125 mg/dL The diagnosis will be based on two abnormal test results, for FBG or RBG and HbA1c, from the same sample or in two separate test samples.
  Interventions: Radiation: Cardiac catheterization
- Normal glycemia: HbA1c <5.7% and FBG 110 mg/dL
  Interventions: Radiation: Cardiac catheterization

INTERVENTIONS:
Radiation: Cardiac catheterization — All the study population will be exposed to diagnostic coronary angiography and invasive coronary intervention as per standard guidelines.

SUMMARY:
This cohort study will measure how severe is the coronary artery disease (CAD), at time of CAD diagnosis, clinically and angiographically in the different cohorts of newly diagnosed diabetes and prediabetes versus normal glycemia patients in the study center.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with consents.
* First time diagnosis of CAD and no prior diagnosis of diabetes milletus (DM), or prediabetes.
* Coronary artery disease confirmed by invasive coronary angiography.

Exclusion Criteria:

1. Patients with known significant anemia, increased hemoglobin turnover, active hemoglobin drops or on erythropoietin therapy.
2. Pregnant and post-partum patients (up to 3 months post-delivery).
3. Patients with severe chronic renal failure (estimated glomerular filtration rate (eGFR) < 30 mL/min/1.72 m2).
4. Patients on any medications with glucose lowering effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A single center cohort study, where all comers, adult patients without prior diagnosis of DM, who are admitted with a first-time diagnosis of CAD, as confirmed by invasive coronary angiography, either elective or as emergency, will be eligible. The study will prospectively enroll consecutives and contemporary cases for each group of diabetes, pre-diabetes and normal glycemia.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease severity | 1 day (During the hospital admission)
  To measure how severe is the CAD, at time of CAD diagnosis, clinically and angiographically in the different cohorts of newly diagnosed diabetes and prediabetes versus normal glycemia patients.

SECONDARY OUTCOMES:
Correlation of HbA1c to CAD severity | 1 day (During the hospital admission)
  To correlate the level of HbA1c to the clinical and angiographic severity of CAD in the study populations

CONTACTS AND LOCATIONS:
Locations (1):
- Saud Albatain cardiac Center, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No